CLINICAL TRIAL: NCT00021034
Title: Phase I Trial of Taurolidine After Positive Second Look Surgery for Recurrent Ovarian Epithelial, Fallopian Tube and Primary Peritoneal Cancers
Brief Title: Taurolidine in Treating Patients With Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-020; CDR0000068740 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1976
Record Dates: First submitted 2001-07-11; First posted 2004-02-16 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Drug Therapy; taurolidine

INTERVENTIONS:
Drug: chemotherapy
Drug: taurolidine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of taurolidine in treating patients who have recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and recommended phase II dose of taurolidine after positive second-look surgery in patients with recurrent ovarian, fallopian tube, or primary peritoneal cancer. II. Determine the dose-limiting toxicity and safety of this drug in these patients.

OUTLINE: This is a dose-escalation study. Patients receive taurolidine intraperitoneally weekly on weeks 1-3 and 7-9 in the absence of disease progression or unacceptable toxicity. Cohorts of 1-6 patients receive escalating doses of taurolidine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Patients are followed every 3 weeks for 9 weeks.

PROJECTED ACCRUAL: A maximum of 15 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal adenocarcinoma Stage IIC or higher at diagnosis Successfully received prior chemotherapy Undergone initial cytoreductive surgery Evidence of gross disease at second-look surgery

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST and/or ALT less than 3 times upper limit of normal No clinically significant PT/PTT abnormality Renal: Creatinine less than 1.7 mg/dL Other: No known hypersensitivity to taurolidine or its excipients No other clinically significant disease that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics Other: At least 30 days since prior investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States